CLINICAL TRIAL: NCT06210204
Title: Improving Access to Surgical Care: Safety, Efficacy, and Satisfaction With Postoperative Telehealth
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Edward Jones, Deputy Chief of Surgery, VA Eastern Colorado Health Care System
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SDR 24-021-1
Record Dates: First submitted 2023-12-11; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Surgery
Keywords: telehealth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-Person (No Intervention): Patients will follow-up in-person after surgery
- Telehealth (Experimental): Patients will follow-up via phone after surgery
  Interventions: Other: Telehealth follow-up

INTERVENTIONS:
Other: Telehealth follow-up — Patients to follow-up via phone after surgery
  Arms: Telehealth

SUMMARY:
Background: A quarter of US Veterans reside in rural communities and are significantly older than their urban counterparts. Providing timely access to care is especially important in this older, independent and medically complex cohort. Virtual care, by phone or video, has improved access to care in non-surgical specialties; however, its utilization in surgery is less than 10% and has continued to decline after the COVID pandemic. Recent studies in surgical patients have demonstrated no difference in missed adverse events, emergency department visits or readmissions; but these data are limited to routine, low-risk procedures in large, urban centers. Routine telehealth for low and high-complexity surgery could be of particular benefit to rural patients by reducing travel challenges, costs, improving scheduling flexibility and reinforcing independence. The hypothesis is that routine telehealth follow-up for elective surgical procedures, of all complexity, will provide equivalent outcomes and improved patient satisfaction and access in comparison to face-to-face follow-up.

Significance: VA Integrated Service Network (VISN) 19 is the largest geographic region in the VA system and includes four intermediate/complex VA Medical Centers (VAMC) serving rural and urban patients across 10 states. Almost 4000 unique patients are seen annually at these 4 centers resulting in 2600 operations and over 16,000 patient encounters. Another 2500 unique patients are referred to community care (CC) at a cost of over $5 million in FY23. Improving access through telehealth in this largely rural VISN will positively impact Veterans and reduce community care expenditures in addition to improving patient and provider satisfaction.

Innovation & Impact: There are currently no funded or published randomized trials evaluating the efficacy of telehealth in providing postoperative surgical care to rural patients. The proposal will provide robust, Level 1 data confirming the safety of postoperative telehealth care. In addition, the investigators will provide the only evaluation of both the patient and provider experience in rural, surgical telehealth care. They will leverage the largest geographic region, VISN19, to ensure broad applicability of findings to rural and urban Veterans.

Specific Aims: Aim 1: Evaluate the safety of postoperative telehealth in rural and urban Veterans. Aim 2: Evaluate the usability and patient satisfaction of telehealth in comparison to in-person postoperative follow-up. Aim 3: Evaluate the usability and provider satisfaction of telehealth in comparison to in-person follow-up.

Methodology: Patients undergoing elective general surgical procedures (both inpatient and outpatient) at four VA medical centers (Denver, CO; Oklahoma City, OK; Muskogee, OK; Salt Lake City, UT) in VISN 19 will be randomized to post-operative follow-up in person or via telehealth. Patients who discharge with drains or wound vacuum therapy, permanent suture or staples will be excluded. Aim 1: 30-day morbidity, missed adverse events (complications that may have been recognized with in-person follow-up), 30-day mortality, 30-day readmission, and 30-day ED visits will be compared evaluated to determine safety of telehealth follow-up. Aim 2: Post-operative surveys at 6 weeks after surgery will quantify acceptability of telehealth follow-up via the standardized Telehealth Usability Questionnaire; satisfaction and usability will be compared via the Consumer Assessment of Healthcare Providers and Systems Outpatient and Ambulatory Surgery survey (S-CAHPS) between the groups. Patients will also be characterized by baseline demographics, distance to nearest facility, socioeconomic vulnerability and procedure type to further define optimal cohorts for future telehealth participation and implementation. Aim 3: Usability and satisfaction for Providers will be determined by self-developed survey. Bi-monthly responses will be recorded to define trends and optimize future implementation.

Next Steps/Implementation: If safe and acceptable to patients and providers, standardization for telehealth follow-up after surgery can be implemented nation-wide to improve access to care and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing general surgery or surgical oncologic surgeries

Exclusion Criteria:

* patients with placement of permanent sutures, wound vacuum devices, staples or other wound devices or drains that would require in-person postoperative follow-up for removal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Missed Adverse Events | 30 days
  Complications that could have been identified with routine follow-up
Patient Satisfaction | 6 weeks
  5-point Likert Scale
Provider Satisfaction | 6 weeks
  5-Point Likert Scale

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Rocky Mountain Regional VAMC, Aurora, Colorado
  - Eastern Oklahoma VAMC, Muskogee, Oklahoma
  - Oklahoma CIty VAMC, Oklahoma City, Oklahoma
  - Salt Lake City VAMC, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
Given the multiple site locations, we are unable to share data without sharing information that can be used to identify individual Veterans and VA Medical Centers.